CLINICAL TRIAL: NCT01981746
Title: Adductor Canal Block and Effect of 10 Versus 30 ml Ropivacaine on Muscle Strength: a Randomized Study in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-PJ-13
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Muscle Strength; Healthy Volunteers
Keywords: adductor canal block; healthy volunteers; US-guided peripheral nerve block; lower limb

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 ml (Experimental): 30 ml ropivacaine 0.1%, single bolus
  Interventions: Procedure: Adductor canal block with ropivacaine 0.1%
- 10 ml (Experimental): 10 ml 0.1% ropivacaine, single bolus
  Interventions: Procedure: Adductor canal block with ropivacaine 0.1%

INTERVENTIONS:
Procedure: Adductor canal block with ropivacaine 0.1% — US-guided adductor canal block

SUMMARY:
To investigate whether reducing the volume (30 versus 10 ml) ropivacaine injected can reduce the number of subjects with impaired muscle strength following adductor canal block. We hypothesized that adductor canal block with 10 ml 0.1% ropivacaine preserves quadriceps strength compared with an adductor canal block with 30 ml.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Men
* ASA 1
* Body Mass Index 18-25

Exclusion Criteria:

* Allergy to study medication
* Earlier trauma or surgery to the lower limb
* Diabetes Mellitus

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with reduced quadriceps strength | 0.5 to 6 hours post block
  The difference between the two volumes in number of subjects experiencing a reduction in quadriceps muscle strength by more than 25% from baseline in two consecutive assessments.

SECONDARY OUTCOMES:
Quadriceps strength in percentage of baseline | 2, 3 and 4 hours post block
  The difference between the two volumes in maximum voluntary isometric contraction (MVIC) of the quadriceps muscle, assessed as percentage of the baseline value.
Quadriceps strength calculated as AUC | 30 minutes to 6 hours post block
  The difference between the two volumes in maximum voluntary isometric contraction (MVIC) of the quadriceps muscle calculated as "area under the curve" (AUC)
Modified 30-second Chair Stand test | 2 and 4 hours post block
  The difference between the pre block value and the post block value in the modified 30-second Chair Stand test performed on one leg, between the two volumes.
VAS pain scores during warmth stimulation | Mean value for the periode 30 minutes - 6 hours post block
  The difference between the two volumes in VAS pain score during warmth stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jaeger, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Jaeger P, Grevstad U, Koscielniak-Nielsen ZJ, Sauter AR, Sorensen JK, Dahl JB. Does dexamethasone have a perineural mechanism of action? A paired, blinded, randomized, controlled study in healthy volunteers. Br J Anaesth. 2016 Nov;117(5):635-641. doi: 10.1093/bja/aew318. PMID 27799178
- [Derived] Jaeger P, Koscielniak-Nielsen ZJ, Hilsted KL, Fabritius ML, Dahl JB. Adductor Canal Block With 10 mL Versus 30 mL Local Anesthetics and Quadriceps Strength: A Paired, Blinded, Randomized Study in Healthy Volunteers. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):553-8. doi: 10.1097/AAP.0000000000000298. PMID 26237001